CLINICAL TRIAL: NCT01553318
Title: Novel Use of Ketotifen (Mast Cell Stabilizer) in Fibromyalgia: A Pilot Study
Brief Title: Novel Use of (Oral) Ketotifen for the Treatment of Fibromyalgia: A Pilot Study
Acronym: KetoforFMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1106005839 (1106-01)
Record Dates: First submitted 2012-03-01; First posted 2012-03-14 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; FMS
MeSH Terms: conditions — Fibromyalgia | interventions — Ketotifen; ketotifen fumarate ophthalmic solution; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Ketotifen (Active Comparator): After meeting the full eligibility requirement, participants will be randomized. Approximately 26 of the 51 participants will assigned to this arm of the study.
  Interventions: Drug: Ketotifen
- Placebo for Ketotifen (Placebo Comparator): After meeting the full eligibility requirement, participants will be randomized. Approximately 25 of the 51 participants will assigned to this arm of the study. Subjects in this arm will receive the placebo drug.
  Interventions: Drug: Placebo (Sugar Pill)

INTERVENTIONS:
Drug: Ketotifen — After meeting the full eligibility requirement, participants will be randomized. From week 1 to 2, subjects will receive either ketotifen 1 mg by mouth, twice a day or the equivalent placebo. Thereafter, subjects will take ketotifen to 2 mg by mouth twice a day or the equivalent placebo.
  Other Names: Zaditor
  Arms: Active Ketotifen
Drug: Placebo (Sugar Pill) — After meeting the full eligibility requirement, participants will be randomized. From week 1 to 2, subjects will receive either ketotifen 1 mg BID or the equivalent placebo. Thereafter, subjects will take ketotifen to 2 mg BID or the equivalent placebo.
  Other Names: Placebo; Sugar Pill
  Arms: Placebo for Ketotifen

SUMMARY:
The purpose of this 10-week study is to determine the effects of a medication called Ketotifen on pain sensitivity; and fibromyalgia-related pain.

Ketotifen works by inhibiting (to prevent or slow down) certain substances in the body that are known to cause inflammation. It is an antihistamine that reduces the harmful effects of histamine. The ophthalmic (eye drops) formulation of ketotifen has been approved by the Food and Drug Administration (FDA) and has been available in the United States for more than a decade. Oral (taken by mouth) ketotifen has been in available in other countries for several decades. Commonly prescribed for the maintenance treatment of asthma and allergic rhinitis, ketotifen has long track record of safety. To date, the oral form of ketotifen has not been approved by the FDA, therefore this study is referred to as an "investigational drug study." Prior to opening recruitment an "investigational new drug" (IND) application which included scientific data and information regarding human safety plans was submitted to and approved by the FDA.

DETAILED DESCRIPTION:
Approximately 46 subjects will be participating in this research. Each subject will be randomized (like flipping a coin) to one of two groups; approximately 23 volunteers will be randomized to receive the active medication and 23 will receive the placebo. Both groups will be "blinded" (will not know) to which group they have been assigned.

The study will be conducted at the Indiana University Clinical Research Center for Pain (CRCP), located on the IUPUI campus in the National Institute of Fitness and Sport building,at 250 University Blvd.,Suite 118 Indianapolis, Indiana, 46202.

To summarize: The subject will be asked to visit the CRCP on four separate occasions: Initial Screening, Week 1, Week 2, and Week 10. This study also includes, answering questionnaires, taking study medication, maintaining a written medication diary and agreeing to remain in weekly contact with the study team to answer a short side effect questionnaire. The side effect questionnaire will be conducted from week 1-4 and then once every 2 weeks from week 4-10.

Study Overview:

Week 0 (clinic visit 1):

1. Informed consent and initial screening questionnaire,
2. Review of all current medications
3. Light physical assessment, e.g. blood pressure, height, weight
4. The investigators will obtain a urine sample for a urine pregnancy test (UPT)
5. Complete short thumb pressure testing in order to set the testing parameters for futures tests (week 1 and week 10)
6. Receive 'pain score' wrist monitor with instructions to record his/her pain level three times each day for one week
7. Receive a one-week medication packet along with instructions to take one tablet twice a day for seven days along with entering dosing information in a medication diary.

Week 1 (clinic visit 2):

1. Submit his/her pain score wrist monitor
2. Submit his/her medication diary for review and return any unused medication
3. Complete the self-assessment questionnaires via computer
4. Undergo a thumb pressures pain sensitivity test
5. If qualified to continue, the subject will receive the next 7-day supply of either a placebo or the active medication, ketotifen 1 mg. along with verbal and written instructions and a medication diary.

Week 2 (visit 3):

1. The investigators will assess the subject's willingness to continue study participation.
2. Review medication diary and medication side-effect/benefit checklist along with any unused study medication. If the subject has not experienced any bothersome side effect and agree to continue,he/she will be issued the next level of either the placebo or the active medication Ketotifen (2 mg.).
3. To assure the subjects' safety, the project coordinator or a member of the research team will complete a medication side-effect questionnaire. The subject will be asked to schedule a weekly check-in call for week 3 and 4 and once every 2 weeks from week 4 to week 10 (weeks 6, 8, and 10)

Week 10 (visit 4):

1. One week prior to this visit, the subject will receive a 'pain score' wrist monitor via an express delivery service (e.g., FedEx) and will be asked to enter his/her pain level three times a day for one week. Then return it during this visit.
2. Review medication side effect/benefit checklist, medication diary and return any unused medication.
3. Completion of self-assessment questionnaires via computer
4. Undergo a thumb pressures pain sensitivity test.

ELIGIBILITY:
Inclusion Criteria:

In order to qualify the subject:

1. must have been diagnosed with fibromyalgia by a medical doctor
2. must be between the ages of 18 to 65 years of age
3. must have a weekly overall body pain average score ≥ 4
4. must pass a screening questionnaire that calculates a physical impairment of ≥ 10
5. must be on stable doses of his/her current medication for at least past four weeks
6. must limit any changes in his/her medication(s) (e.g., dose change, addition or discontinuation of any medication that effects the central nervous system, e.g., benzodiazepines, sedative/hypnotic, etc. ) during the 10-week study period unless medically necessary
7. must report all medication including herbal supplements and over-the-counter medications, e.g. cold medication, eye drops, etc. that he/she is currently taking to a member of the research team
8. must be willing to maintain a medication diary provided to him/her during the 10-week study period
9. must be willing to abstain (not take) any fibromyalgia related medication including over-the-counter for at least 8-hours prior to each of the two testing visits (Otherwise, he/she may take these medication(s) immediately after pain sensitivity testing has been completed and as prescribed in-between visits)
10. must agree to use a proven method of contraception to prevent pregnancy throughout this study

Exclusion Criteria:

The subject will not be allowed to participate if:

1. he/she has a history of seizures
2. he/she has atopic dermatitis (also called eczema) or chronic urticaria (hives)
3. he/she has chronic thrombocytopenia (a low blood platelet count)
4. she is currently pregnant, are planning to become pregnant, or is breastfeeding
5. he/she has been diagnosed by a psychiatrist with Schizophrenia or bipolar disorder
6. he/she has been diagnosed with another major rheumatic conditions (i.e. rheumatoid arthritis, systemic lupus erythematosus, scleroderma and/or other connective tissue diseases)
7. he/she plans to undergo an elective surgery within the study timeline
8. he/she is in the process of filing, or plan to file for disability benefits within the study timeline
9. his/her screening labs results are abnormal (i.e., elevated SGPT and low platelet count)
10. he/she is currently using any anti-allergy drugs (ophthalmic or oral histamine antagonist), leukotriene inhibitors (e.g., montelukast) or prednisone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis C. Ang, MD, Principal Investigator — Wake Forest University
Locations (1):
- IU Clincial Research Center for Pain and Fibromyalgia, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketotifen: ketotifen active group
- Placebo: Placebo medication
Period: Overall Study
Arm/Group | Ketotifen | Placebo
Started | 24 | 27
Completed | 21 | 25
Not Completed | 3 | 2
Not completed — Protocol Violation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ketotifen Group: Participants who received the active drug - ketotifen
- Placebo: Participants who received the placebo
- Total: Total of all reporting groups
Arm/Group | Ketotifen Group | Placebo | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (8.5) | 51.3 (8.5) | 51.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51
weekly average pain score [Mean (Standard Deviation); unit: units on a scale] — Average of daily pain scores within a one week period (scale from 0 to 10, with 10 being the worse pain possible)
  units on a scale | 6.5 (0.9) | 6.2 (1.3) | 6.4 (1.1)
Fibromyalgia impact questionnaire [Mean (Standard Deviation); unit: units on a scale] — Score range from 0 to 100 with higher scores indicating worse health status
  units on a scale | 66.9 (16.2) | 66.6 (12.0) | 66.8 (14.0)
Evoked pain [Mean (Standard Deviation); unit: units on a scale] — Range from 0 to 20, with higher score representing greater sensitivity to pressure pain stimuli
  units on a scale | 10.3 (0.4) | 9.8 (0.4) | 10.0 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Average Pain Score on the Visual Analog Scale at Week 10
Description: Change in weekly average pain score from baseline to week 10 (range from -10 to +10): interpretation= the more negative the value is, the larger reduction in pain severity at week 10 is
Time Frame: baseline and week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketotifen: Ketotifen active drug
- Placebo: received placebo
Arm/Group | Ketotifen | Placebo
Number analyzed (Participants) | 24 | 27
units on a scale | -1.33 (1.92) | -1.54 (1.93)

2. Secondary Outcome: Change From Baseline in Evoked Pain Score at Week 10
Description: Change in evoked pain score from baseline to week 10 (scale range -20 to +20): interpretation= the more negative the value is, the larger the reduction in sensitivity to pressure pain stimuli
Time Frame: baseline and week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketotifen: active drug group
- Placebo: placebo group
Arm/Group | Ketotifen | Placebo
Number analyzed (Participants) | 24 | 27
units on a scale | -0.33 (0.36) | -0.27 (0.34)

3. Secondary Outcome: Fibromyalgia Impact Questionnaire
Description: Change in global symptom severity [scale range from -100 to +100] = the more negative the value is, the greater the improvement in overall symptom severity
Time Frame: baseline and week 10
Population: Indeed, fibromyalgia impact questionnaire is a secondary outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketotifen | Placebo
Number analyzed (Participants) | 24 | 27
units on a scale | -12.13 (19.54) | -12.27 (18.12)

4. Secondary Outcome: Change From Baseline in the Blood Levels of IL-8, MCP-1 and Eotaxin at Week 10
Description: Change in peripheral blood levels of IL-8, MCP-1 and Eotaxin from baseline to week 10
Time Frame: baseline and week10
Population: We do not have data on the chemokines because of the problems we had with the assays. Indeed, IL-8, MCP-1 and Eotaxin were all secondary outcomes.
Arm/Group | Ketotifen | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Ketotifen: Received ketotifen the active drug
Arm/Group | Ketotifen | Placebo
Serious Adverse Events (participants affected / at risk) | 6/24 | 1/27
Other Adverse Events (participants affected / at risk) | 3/24 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketotifen (N=24) | Placebo (N=27)
transient drowsiness (Nervous system disorders) | 6 (6) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketotifen (N=24) | Placebo (N=27)
Fatigue (Psychiatric disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Just tested one dose (low dose). Would be better if we tested higher dosages

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No